CLINICAL TRIAL: NCT01880463
Title: Dry Eye Disease in the Vitamin D and Omega-3 Trial (VITAL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Debra Ann Schaumberg, ScD, OD, MPH, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012P001332; R01EY022663 (NIH)
Record Dates: First submitted 2013-06-15; First posted 2013-06-19 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Dry Eye Disease
Keywords: Dry eye disease; incidence; progression
MeSH Terms: conditions — Dry Eye Syndromes; Disease Progression | interventions — Fatty Acids, Omega-3; Fish Oils; Omacor; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D + fish oil placebo (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day
  Fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3; Drug: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator): Vitamin D placebo
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg. of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3 placebo
- Vitamin D placebo + fish oil placebo (Placebo Comparator): Vitamin D placebo
  fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 placebo; Drug: Fish oil placebo
- Vitamin D + fish oil (Active Comparator): Vitamin D (cholecalciferol), 2000 IU per day
  Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg. of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3

INTERVENTIONS:
Drug: Omega-3 fatty acids (fish oil)
  Other Names: Omacor
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D3
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Dietary Supplement: Vitamin D3 placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Drug: Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 Trial (VITAL; NCT 01169259) is a randomized clinical trial in 25,875 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL and will examine whether omega-3 fatty acids or vitamin D3, compared to placebo, reduce the incidence and/or progression of dry eye disease.

DETAILED DESCRIPTION:
This ancillary study to VITAL will examine the efficacy of omega-3 fatty acids and vitamin D3 in prevention of dry eye disease. The primary aims are to test whether omega-3 fatty acid supplementation (1) reduces the incidence of dry eye disease, and (2) improves the natural history of dry eye disease by relieving symptoms and other impacts on quality of life. Secondary aims are to estimate the incidence of dry eye disease in the US, prospectively examine the natural history of dry disease, explore factors that could modify or influence the impact of omega-3 fatty acid supplementation, evaluate the interrelationship of dry eye disease and depression, and test for possible independent or joint effects of vitamin D3 supplementation in the incidence and natural history of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* All participants in VITAL (NCT 01169259) are eligible to participate in this ancillary study.

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25875 (Actual)
Dates: Start 2010-07; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Dry Eye Disease | 5 years
  Report of a diagnosis of dry eye disease confirmed by medical record review.

REFERENCES:
- [Derived] Christen WG, Cook NR, Manson JE, Buring JE, Lee IM, Bubes V, Friedenberg G, Dushkes R, Smith D, Schaumberg DA; VITAL Research Group. Efficacy of Marine omega-3 Fatty Acid Supplementation vs Placebo in Reducing Incidence of Dry Eye Disease in Healthy US Adults: A Randomized Clinical Trial. JAMA Ophthalmol. 2022 Jul 1;140(7):707-714. doi: 10.1001/jamaophthalmol.2022.1818. PMID 35679030
- See also: Welcome to the VITAL Study website — http://vitalstudy.org